CLINICAL TRIAL: NCT04876261
Title: Bioavailability of Hydroxytyrosol From Two Olive Watery Extract Supplements and Their Effects on Lipid Peroxidation
Brief Title: Bioavailability of Hydroxytyrosol From Olive Watery Extract Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daacro (Network)
Collaborators: ISTITUTO KURZ ITALIA S.R.L. (Unknown); Institut Kurz GmbH (Unknown); Fattoria La Vialla di Gianni, Antonio e Bandino Lo Franco Soc. Agr. Sempl. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IK03-2020
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Biological Availability
Keywords: Olives
MeSH Terms: interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Intervention Model Description: Three-armed study with a cross-over design. Participants will be randomly assigned to either group A, B or C. The group allocation will define the sequence of product intake:
  * Group A: first OliPhenolia® bitter, second OliPhenolia®, third La Vialla Extra Virgin Olive Oil
  * Group B: first OliPhenolia®, second La Vialla Extra Virgin Olive Oil, third OliPhenolia® bitter
  * Group C: first La Vialla Extra Virgin Olive Oil, second OliPhenolia® bitter, third OliPhenolia®
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the laboratory will be blinded. Laboratory staff will be unblinded after samples are being analysed. Participants will be unblinded after study end.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Group A will receive Oliphenolia® bitter on intervention visit 1 followed by Oliphenolia® on intervention visit 2 and followed by La Vialla Extra Virgin Olive Oil with 5 mg hydroxytyrosol on the third and final intervention visit
  Interventions: Dietary Supplement: Oliphenolia® bitter; Dietary Supplement: Oliphenolia®; Dietary Supplement: La Vialla Extra Virgin Olive Oil containing 5 mg hydroxytyrosol
- Group B (Active Comparator): Group B will receive Oliphenolia® on intervention visit 1 followed by La Vialla Extra Virgin Olive Oil with 5 mg hydroxytyrosol on intervention visit 2 and followed by Oliphenolia® bitter on the third and final intervention visit
  Interventions: Dietary Supplement: Oliphenolia® bitter; Dietary Supplement: Oliphenolia®; Dietary Supplement: La Vialla Extra Virgin Olive Oil containing 5 mg hydroxytyrosol
- Group C (Active Comparator): Group C will receive La Vialla Extra Virgin Olive Oil with 5 mg hydroxytyrosol on intervention visit 1 followed by Oliphenolia® bitter on intervention visit 2 and followed by Oliphenolia® on the third and final intervention visit
  Interventions: Dietary Supplement: Oliphenolia® bitter; Dietary Supplement: Oliphenolia®; Dietary Supplement: La Vialla Extra Virgin Olive Oil containing 5 mg hydroxytyrosol

INTERVENTIONS:
Dietary Supplement: Oliphenolia® bitter — * ingredients: concentrated watery extract of olives 94%, lemon juice 6%
  * 35 mg hydroxytyrosol, 0,24 mg Oleuropein
Dietary Supplement: Oliphenolia® — * ingredients: grape juice concentrate 70%, concentrated watery extract of olives 30%
  * 38 mg hydroxytyrosol, 0,28 mg Oleuropein
Dietary Supplement: La Vialla Extra Virgin Olive Oil containing 5 mg hydroxytyrosol — * extra virgin olive oil
  * 5 mg hydroxytyrosol

SUMMARY:
The aim of this cross-over study is to assess the bioavailability of hydroxytyrosol in healthy males after the intake of two olive watery extract supplements and one olive oil. Blood and urine samples will be collected before and after intake of the investigational products. Sample will be analysed regarding the level of hydroxytyrosol and preventing lipid peroxidation.

DETAILED DESCRIPTION:
Background:

Hydroxytyrosol is a phenolic phytochemical naturally occurring in olives with potential antioxidant, anti-inflammatory, and health benefits mainly related with cardiovascular diseases [for review see Covas et al., 2015]. OliPhenolia® bitter and OliPhenolia® are two food supplements resulting from the liquid by-product generated during olive oil production, that are rich in olive polyphenols, mainly hydroxytyrosol. Hydroxytyrosol and its derivatives (tyrosol and oleuropein) are present in higher levels in the watery extracts from olives when compared with the oil fraction.

Most studies on hydroxytyrosol bioavailability have been performed by consuming it with olive oil or as a highly purified molecule. In a study by D'Angelo and collaborators [D'Angelo et al, 2001] it was shown that hydroxytyrosol can be rapidly absorbed from the blood and distributed in the human body, metabolized and eliminated rapidly in urine mainly as a glucuronide. It has been estimated that the absorption process depends on the composition of the food matrix through which hydroxytyrosol is administered [Visioli et al, 2003], when consumed together with fats (e.g. olive oil) it is absorbed in a greater extent. By being a water-soluble molecule, hydroxytyrosol is only slightly soluble in fats, therefore naturally present in significantly higher concentrations in the olive fruit aqueous fractions than in the olive oil.

Overall, the human studies support the need to evaluate the bioavailability of hydroxytyrosol following its administration as a major component of the two aqueous food supplements, OliPhenolia® and OliPhenolia® bitter.

Study Procedure:

After detailed information and signed informed consent all males meeting the inclusion and exclusion criteria will be included into the study. During their study participation, participants are not allowed to consume any products with or made from olives or olive oil as well as alcohol and supplements with hydroxytyrosol, vitamins, minerals and antioxidants. Products high in polyphenols and antioxidants may only be consumed in moderate amounts. Three days prior to and at each intervention day, volunteers will be requested to avoid moderate or intense physical activity.

After a run-in period, participants will return in a fasted state to the site for the first intervention visit. Volunteers will be asked to empty their bladder at home 2h before IP intake. After arriving at the site, a baseline blood and urine sample (-5 min) will be collected and the participants receive according to the individual allocation determining the sequence of the IP intake either one of the olive watery extract supplements (OliPhenolia® bitter or OliPhenolia®) or the olive oil first. Further blood and urine samples will follow (+30 min, +60 min, +90 min, +120 min, +240 min, +12 h). Vital signs and AEs will be checked throughout the intervention visit. Participants will receive several snacks and water during their visit.

After a one-week washout phase each, participants will return to their second and third intervention visit. The same procedures as on intervention visit 1 will take place except the IP intake will vary according to the individual allocation.

At the end of the third intervention visit, participants will receive a study compensation.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy men aged 21-50,
* subject has an adequate understanding of the study and signs the informed consent to participate in the study,
* willingness to follow dietary and physical activity restrictions during study participation,
* body mass index range: >18.5 and <29.9 kg/m2.

Exclusion Criteria:

* Any known allergies to IPs (olives and their derivates),
* any acute and chronic diseases (e.g. diagnosis of diabetes mellitus, hypertension, dyslipidemia or other cardiometabolic disorders, diagnosed hepatic, renal, or cardiovascular disease),
* any kind of eating disorders,
* not fluent in German,
* any previous (last 14 days prior to screening) and any ongoing pharmacological therapy (e.g. any medication, vaccination, infusion),
* any intake of nutritional supplements,
* any known addiction to drugs and/or alcohol,
* smoker,
* Investigator or physician doubts truthfulness of self-reported health information.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability of hydroxytyrosol in urine | -2 hrs to IP intake, 0 to 30 min, 30 to 60 min, 60 to 90 min, 90 to 120 min, 120 to 240 min and +4h to +12h
  The primary objective is the bioavailability of hydroxytyrosol and its derivatives from both food supplements (OliPhenolia® bitter and OliPhenolia®) in urine when compared to extra virgin olive oil.
Bioavailability of hydroxytyrosol in blood | 5 min. before IP intake, 30, 60, 90, 120, 240 min and 12 h
  The primary objective is the bioavailability of hydroxytyrosol and its derivatives from both food supplements (OliPhenolia® bitter and OliPhenolia®) in urine when compared to extra virgin olive oil.

SECONDARY OUTCOMES:
Oxidative damages to lipids in blood | 5 min. before IP intake, 30, 60, 90, 120, 240 min and 12 h
  The secondary outcome is the measurement of the oxidized LDL(low-density lipoprotein) in blood
changes in F2alpha-isoprostanes in urine | -2 hrs to IP intake, 0 to 30 min, 30 to 60 min, 60 to 90 min, 90 to 120 min, 120 to 240 min and +4h to +12h
  The secondary outcome is the measurement of changes in F2alpha-isoprostanes in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, PhD, Principal Investigator — Daacro
Locations (1):
- daacro GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Angelo S, Manna C, Migliardi V, Mazzoni O, Morrica P, Capasso G, Pontoni G, Galletti P, Zappia V. Pharmacokinetics and metabolism of hydroxytyrosol, a natural antioxidant from olive oil. Drug Metab Dispos. 2001 Nov;29(11):1492-8. PMID 11602527
- [Background] Caruso D, Visioli F, Patelli R, Galli C, Galli G. Urinary excretion of olive oil phenols and their metabolites in humans. Metabolism. 2001 Dec;50(12):1426-8. doi: 10.1053/meta.2001.28073. PMID 11735087
- [Background] Covas MI, Nyyssonen K, Poulsen HE, Kaikkonen J, Zunft HJ, Kiesewetter H, Gaddi A, de la Torre R, Mursu J, Baumler H, Nascetti S, Salonen JT, Fito M, Virtanen J, Marrugat J; EUROLIVE Study Group. The effect of polyphenols in olive oil on heart disease risk factors: a randomized trial. Ann Intern Med. 2006 Sep 5;145(5):333-41. doi: 10.7326/0003-4819-145-5-200609050-00006. PMID 16954359
- [Background] Covas MI, de la Torre R, Fito M. Virgin olive oil: a key food for cardiovascular risk protection. Br J Nutr. 2015 Apr;113 Suppl 2:S19-28. doi: 10.1017/S0007114515000136. PMID 26148918
- [Background] de Bock M, Thorstensen EB, Derraik JG, Henderson HV, Hofman PL, Cutfield WS. Human absorption and metabolism of oleuropein and hydroxytyrosol ingested as olive (Olea europaea L.) leaf extract. Mol Nutr Food Res. 2013 Nov;57(11):2079-85. doi: 10.1002/mnfr.201200795. Epub 2013 Jun 14. PMID 23766098
- [Background] Hohmann CD, Cramer H, Michalsen A, Kessler C, Steckhan N, Choi K, Dobos G. Effects of high phenolic olive oil on cardiovascular risk factors: A systematic review and meta-analysis. Phytomedicine. 2015 Jun 1;22(6):631-40. doi: 10.1016/j.phymed.2015.03.019. Epub 2015 Apr 20. PMID 26055128
- [Background] Karkovic Markovic A, Toric J, Barbaric M, Jakobusic Brala C. Hydroxytyrosol, Tyrosol and Derivatives and Their Potential Effects on Human Health. Molecules. 2019 May 24;24(10):2001. doi: 10.3390/molecules24102001. PMID 31137753
- [Background] Mateos R, Martinez-Lopez S, Baeza Arevalo G, Amigo-Benavent M, Sarria B, Bravo-Clemente L. Hydroxytyrosol in functional hydroxytyrosol-enriched biscuits is highly bioavailable and decreases oxidised low density lipoprotein levels in humans. Food Chem. 2016 Aug 15;205:248-56. doi: 10.1016/j.foodchem.2016.03.011. Epub 2016 Mar 4. PMID 27006237
- [Background] Miro-Casas E, Covas MI, Fito M, Farre-Albadalejo M, Marrugat J, de la Torre R. Tyrosol and hydroxytyrosol are absorbed from moderate and sustained doses of virgin olive oil in humans. Eur J Clin Nutr. 2003 Jan;57(1):186-90. doi: 10.1038/sj.ejcn.1601532. PMID 12548315
- [Background] Suarez M, Valls RM, Romero MP, Macia A, Fernandez S, Giralt M, Sola R, Motilva MJ. Bioavailability of phenols from a phenol-enriched olive oil. Br J Nutr. 2011 Dec;106(11):1691-701. doi: 10.1017/S0007114511002200. Epub 2011 Jun 21. PMID 21736768
- [Background] Visioli F, Galli C, Bornet F, Mattei A, Patelli R, Galli G, Caruso D. Olive oil phenolics are dose-dependently absorbed in humans. FEBS Lett. 2000 Feb 25;468(2-3):159-60. doi: 10.1016/s0014-5793(00)01216-3. PMID 10692578
- [Background] Visioli F, Galli C, Grande S, Colonnelli K, Patelli C, Galli G, Caruso D. Hydroxytyrosol excretion differs between rats and humans and depends on the vehicle of administration. J Nutr. 2003 Aug;133(8):2612-5. doi: 10.1093/jn/133.8.2612. PMID 12888646